CLINICAL TRIAL: NCT03208933
Title: Local Open-label Multicenter Study to Assess the Effectiveness of Pirfenidone in Patients With Idiopathic Pulmonary Fibrosis in Russian Clinical Practice
Brief Title: Open-label Study to Assess the Effectiveness of Pirfenidone in Participants With Idiopathic Pulmonary Fibrosis (IPF).
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML39355
Record Dates: First submitted 2017-06-26; First posted 2017-07-06 (Actual); Results first posted 2020-11-20 (Actual); Last update posted 2020-11-20 (Actual); Status verified 2020-11

CONDITIONS: Idiopathic Pulmonary Fibrosis
Keywords: Pirfenidone, UIP, IPF, FVC
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis | interventions — pirfenidone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Pirfenidone (Experimental): Participants will be administered pirfenidone 2403 milligram per day (mg/d) orally for 26 weeks in participants with IPF.
  Interventions: Drug: Pirfenidone

INTERVENTIONS:
Drug: Pirfenidone — Pirfenidone 2403 mg/d capsules orally will be given in divided doses (TID) after titration period of 14 days.
  Other Names: Esbriet, RO0220912

SUMMARY:
This study is a national, multicenter, interventional, non-randomized, non-controlled, open-label study to assess the effectiveness of pirfenidone in participants with IPF in Russian clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Clinical symptoms consistent with IPF of ≥ 6months duration
* Participants could have both "confident" or "consistent" with UIP diagnosis of IPF based on clinical, radiologic and pathologic data according to 2011 American Thoracic Society/European Respiratory Society (ATS/ERS) guidelines at the Screening. HRCT scan performed within 24 months before the start of the Screening may be used, if it meets all image acquisition guideline
* No features supporting an alternative diagnosis on transbronchial biopsy, bronchoalveolar lavage (BAL), or surgical lung biopsy, if performed. Results of the surgical lung biopsy performed within the last 4 years must be confirmed by central review
* Participants with %FVC ≥ 40 % at the Screening
* Participants with %Carbon monoxide diffusing capacity (DLCO) ≥ 30 % at the Screening
* Ability to walk ≥ 100 m during the 6-minute walk test at the Screening
* Eligible participants must discontinue all prohibited medications at least 28 days before the Screening
* Female participants of childbearing potential must have negative urine pregnancy test at the Screening and before first dosing on Day 1

Exclusion Criteria:

* Significant clinical worsening of IPF between Screening and Day 1, in the opinion of the investigator
* Relevant airways obstruction (i.e. pre-bronchodilator forced expiratory volume (FEV)1/FVC < 0.7)
* Cigarette smoking within 28 days before the start of treatment or unwilling to avoid tobacco products throughout the study
* History of clinically significant environmental exposure known to cause pulmonary fibrosis (PF), including but not limited to drugs (such as amiodarone), asbestos, beryllium, radiation, and domestic birds
* Known explanation for interstitial lung disease, including but not limited to radiation, drug toxicity, sarcoidosis, hypersensitivity pneumonitis, bronchiolitis obliterans organizing pneumonia, human immunodeficiency virus (HIV), viral hepatitis, and cancer
* Clinical diagnosis of any connective tissue disease, including but not limited to scleroderma, polymyositis/ dermatomyositis, systemic lupus erythematosus, and rheumatoid arthritis
* During baseline analysis of HRCT, significant coexistent emphysema (emphysema extent greater than extent of fibrosis) confirmed by central review
* Planned lung transplantation during the study
* Clinical evidence of active infection, including but not limited to bronchitis, pneumonia, sinusitis, urinary tract infection, or cellulitis
* Unable to perform 6MWT or to undergo pulmonary function test
* Any history of malignancy likely to result in significant disability or likely to require significant medical or surgical intervention within the next 1 years. This does not include minor surgical procedures for localized cancer (e.g., basal cell carcinoma)
* History of severe hepatic impairment or end-stage liver disease
* History of end-stage renal disease requiring dialysis
* History of unstable or deteriorating cardiac or pulmonary disease (other than IPF) within the previous 6 months
* Pregnancy or lactation, or intention to become pregnant during the study. Women of childbearing capacity are required to have a negative urine pregnancy test before treatment and must agree to maintain highly effective contraception
* Liver function test outside specified limits at the Screening: total bilirubin above the upper limit of normal (ULN); aspartate or alanine aminotransferase (AST or ALT) > 3 × ULN; alkaline phosphatase > 2.5 × ULN
* Creatinine clearance < 30 mL/min, calculated using the Cockcroft-Gault formula
* Electrocardiogram (ECG) with a QT interval corrected according to Fridericia's formula (QTcF) > 500 msec at the Screening

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-10-23 (Actual); Primary Completion 2019-11-13 (Actual); Study Completion 2019-11-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (11):
- Russia (11):
  - Regional State Budgetary Institution of Healthcare "Regional Cinilcal Hospital"; Pulmonology, Barnaul, Altayskiy Kray
  - GBUZ Regional clinical hospital #4, Chelyabinsk, Evenkija
  - Central NII tuberkuleza RAMN, Moscow, Moscow Oblast
  - Pulmonologii NII FMBA of Russia, Moscow, Moscow Oblast
  - SBEI HPE "The First St.Petersburg State Medical University n.a. acad. I.P.Pavlova"of MoH of RF, Saint Petersburg, Sankt-Peterburg
  - New Hospital, Yekaterinburg, Sverdlovsk Oblast
  - I.M. Sechenov First Moscow State Medical University: The E.M. Tareyev Clinic, Moscow
  - Vladimirskiy Regional Scientific Research Inst., Moscow
  - State Novosibirsk Regional Clinical Hospital, Novosibirsk
  - Republican clinical hospital named after G.G. Kuvatov, Ufa
  - Budget Institution of Healthcare of Voronezh Region "Voronezh Regional Clinical Hospital #1", Voronezh

IPD SHARING:
Plan to Share IPD: Yes
CT images of lungs, forced vital capacity (FVC) measurements, post-hoc analysis

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study enrolled participants in Russia.
Groups:
- Pirfenidone: Participants administered pirfenidone 2403 milligram per day (mg/d) orally for 26 weeks
Period: Overall Study
Arm/Group | Pirfenidone
Started | 60
Completed | 47
Not Completed | 13
Not completed — Death | 3
Not completed — Withdrawal by Subject | 3
Not completed — Adverse Event | 1
Not completed — Lost to Follow-up | 2
Not completed — Physician Decision | 3
Not completed — Protocol Violation | 1

BASELINE CHARACTERISTICS:
Arm/Group | Pirfenidone
Number analyzed (Participants) | 60
Age, Continuous [Mean (Standard Deviation); unit: Years] | 67.4 (7.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 41
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Russian | 48
  Tatar | 4
  Bashkir | 4
  Armenian | 1
  Dagestani | 1
  Kazah | 1
  Uzbek | 1

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 26 in Absolute Millilitre (mL) Forced Vital Capacity (FVC)
Description: FVC is a standard pulmonary function test. FVC is defined as the volume of air that can forcibly be blown out after full inspiration in the upright position, measured in liters. Baseline FVC will be the average of the highest FVC measurement recorded at the Screening and Day 1. The FVC at Week 26 will be the average of the highest FVC measurement recorded on two separate days at Week 26.
Time Frame: Baseline, Week 26
Population: Included participants that had data for at least one post-baseline assessment of any efficacy measurement
Measure: Mean (95% Confidence Interval); unit: Milliliter (mL)
Arm/Group | Pirfenidone
Number analyzed (Participants) | 55
Milliliter (mL) | 128.78 [-26.84 to 284.40]

2. Primary Outcome: Change From Baseline to Week 26 in Percent (%) Predicted FVC
Description: Predicted FVC is based on sex, age, and height of a person. Percent predicted FVC (in %) = [(observed FVC)/(predicted FVC)]*100.
Time Frame: Baseline, Week 26
Population: Included participants that had data for at least one post-baseline assessment of any efficacy measurement
Measure: Mean (95% Confidence Interval); unit: percent predicted
Arm/Group | Pirfenidone
Number analyzed (Participants) | 55
percent predicted | -0.10 [-3.18 to 2.99]

3. Secondary Outcome: Change From Baseline to Week 26 in 6-Minute Walk Test (6MWT) Distance
Description: Baseline 6MWT distance will be the average of the measurements recorded at the Screening and Day 1 visits. The 6MWT distance at Week 26 will be defined as the average of the 6MWT distance recorded on two separate days at Week 26.
Time Frame: Baseline, Week 26
Population: Included participants that had data for at least one post-baseline assessment of any efficacy measurement and for the 6MWT at Week 26
Measure: Count of Participants; unit: Participants
Arm/Group | Pirfenidone
Number analyzed (Participants) | 49
Participants
  Decline of >= 50 m | 14
  Decline of <50 m to 0 m | 11
  Improvement of >= 0 m | 24

4. Secondary Outcome: Change From Baseline to Week 26 in EuroQol 5-Dimension 5-Level (EQ-5D-5L) Questionnaire Index Score
Description: The EQ-5D-5L is a self-reported health status questionnaire that consists of six questions used to calculate a health utility score for use in health economic analysis. There are two components to the EQ-5D-5L: a five-item health state profile that assesses mobility, self-care, usual activities, pain/discomfort, and anxiety/depression used to obtain an Index Utility Score, as well as a visual analogue scale (VAS) that measures health state. Overall scores range from 0 to 1, with low scores representing a higher level of dysfunction.
Time Frame: Baseline, Week 26
Population: Included participants that had data for at least one post-baseline assessment of any efficacy measurement
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Pirfenidone
Number analyzed (Participants) | 55
score on scale | -0.0288 (0.1820)

5. Secondary Outcome: Change From Baseline to Week 26 in EQ-5D-5L Visual Analogue Scale (EQ-5D-5L VAS) Score
Description: The EQ-5D-5L is a self-reported health status questionnaire that consists of six questions used to calculate a health utility score for use in health economic analysis. There are two components to the EQ-5D-5L: a five-item health state profile that assesses mobility, self-care, usual activities, pain/discomfort, and anxiety/depression used to obtain an Index Utility Score, as well as a visual analogue scale (VAS) that measures health state. The VAS is designed to rate the participant's current health state on a scale from 0 to 100, where 0 represents the worst imaginable health state and 100 represents the best imaginable health state.
Time Frame: Baseline, Week 26
Population: Included participants that had data for at least one post-baseline assessment of any efficacy measurement
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Pirfenidone
Number analyzed (Participants) | 55
score on scale | -0.6 (17.16)

6. Secondary Outcome: Percentage of Participants With Treatment Emergent Adverse Events (TEAEs) and Treatment Emergent Serious Adverse Events (TESAEs)
Description: An AE is defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (eg, a clinically significant abnormal laboratory finding), symptom, or disease temporally associated with the use of a drug, whether or not it is considered related to the drug. A treatment-emergent adverse event (TEAE) is defined as an adverse event with an onset that occurs after receiving study drug. Serious adverse event is any untoward medical occurrence at any dose that resulted in death, was life-threatening, required inpatient hospitalization or prolongation of hospitalization, or resulted in persistent or significant disability/incapacity or congenital anomaly/birth defect.
Time Frame: Up to Week 52
Measure: Number; unit: percentage of participants
Arm/Group | Pirfenidone
Number analyzed (Participants) | 60
percentage of participants
  TEAEs | 81.7
  TESAEs | 16.7

ADVERSE EVENTS:
Time Frame: Up to 52 Weeks
Arm/Group | Pirfenidone
All-Cause Mortality (participants affected / at risk) | 7/60
Serious Adverse Events (participants affected / at risk) | 10/60
Other Adverse Events (participants affected / at risk) | 32/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pirfenidone (N=60)
Idiopathic pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Death (General disorders) | 2 (2)
Sudden cardiac death (General disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Atrial flutter (Cardiac disorders) | 1 (1)
Bronchitis bacterial (Infections and infestations) | 1 (1)
Cholecystitis infective (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pirfenidone (N=60)
Nausea (Gastrointestinal disorders) | 16
Dyspepsia (Gastrointestinal disorders) | 8
Vomiting (Gastrointestinal disorders) | 8
Diarrhoea (Gastrointestinal disorders) | 7
Decreased appetite (Metabolism and nutrition disorders) | 13
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 4
Weight decreased (Investigations) | 4
Pruritus (Skin and subcutaneous tissue disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights

DOCUMENTS (2):
  • Study Protocol (2019-02-01): https://cdn.clinicaltrials.gov/large-docs/33/NCT03208933/Prot_000.pdf
  • Statistical Analysis Plan (2020-06-17): https://cdn.clinicaltrials.gov/large-docs/33/NCT03208933/SAP_001.pdf